CLINICAL TRIAL: NCT02110316
Title: Bioavailability of Voriconazole in Critically Ill Patients
Brief Title: Bioavailability of Voriconazole
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no eligible patients; study stopped without inclusion
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, JWC Alffenaar, PharmD, PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 47955
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-02

CONDITIONS: Voriconazole; Bioavailability; Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bioavailability (Other): 1 arm, different dosage form
  Interventions: Other: Dosage form of voriconazole

INTERVENTIONS:
Other: Dosage form of voriconazole — Instead of an oral dose of voriconazole, patients receive one intravenous dose of voriconazole (in the same dose as the oral dose).

SUMMARY:
The objective of this study is to obtain the absolute bioavailability of voriconazole in critically ill ICU patients, because pharmacokinetics can be different in critically ill patients due to alterations in function of various organs and body systems compared with healthy volunteers.

DETAILED DESCRIPTION:
The bioavailability of voriconazole, based on healthy volunteers, is estimated to be >90%. Due to the high bioavailability of voriconazole, switching between oral and intravenous administration is permitted if clinically allowed. Few data are available for the bioavailability of voriconazole in critically ill patients. However, to obtain a therapeutic concentration of voriconazole (>1.5 mg/L, which is associated with a beneficial response to treatment) one study showed that a higher oral dose is required compared with the intravenous dose, to obtain this therapeutic concentration. Therefore, the pharmacokinetics can be changed in critically ill patients, including bioavailability.

In this study, patients who receive voriconazole orally (prescribed by their attending physician) will receive one intravenous dose of voriconazole instead of the oral dose. The intravenous dose will be the same as the oral dose voriconazole.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 yrs;
* Treatment with voriconazole;
* Admission to an ICU;
* Written informed consent.

Exclusion Criteria:

* Blood sampling by central venous catheter or peripheral cannula not possible;
* Concomitantly using a strong inhibitor or inducer of cytochrome P450.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The bioavailability of voriconazole in critically ill patients | 1 day
  Bioavailability will be determined by comparing the area under the concentration time curve (AUC) of an intravenous and oral dose of voriconazole.

SECONDARY OUTCOMES:
Correlation of bioavailability of voriconazole with disease severity | 1 day
  Disease severity will be determined using the APACHE IV score
Correlation of bioavailability of voriconazole with the degree of inflammation | 1 day
  To determine the degree of inflammation C-reactive protein (CRP) will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Alffenaar, PharmD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands